CLINICAL TRIAL: NCT01235013
Title: Effect of Maraviroc (MCV) on the Immunological Recovery of HIV-1 Discordant Patients With CD4 Lymphocyte Counts Below 200 Cells/mm3
Acronym: DIS-MVC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Dr. José María Gatell, Hospital Clínic i Provincial de Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DIS-MVC
Record Dates: First submitted 2010-11-04; First posted 2010-11-05 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-10

CONDITIONS: HIV-1 Infection
Keywords: HIV-1 infection; Maraviroc; CD4 lymphocyte count
MeSH Terms: interventions — Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Maraviroc (Experimental)
  Interventions: Drug: Maraviroc
- Control (No Intervention): Patients continue with their usual treatment

INTERVENTIONS:
Drug: Maraviroc — 150 mg of Maraviroc every 12 hours (300 mg daily) orally for 24 weeks
  Arms: Maraviroc

SUMMARY:
Maraviroc is an antiretroviral drug that belongs to the family of the CCR5 coreceptor inhibitors. It has proven to be effective in increasing CD4 lymphocyte counts in both in treated and naïve patients, irrespective of the viral load.

The investigators hypothesize that adding Maraviroc to the antiretroviral treatment of discordant patients, defined as those having CD4 lymphocyte counts below 200 cells /mm3 during the last year, could lead to its immunological recovery.

60 patients will be included in this unicentric, prospective, randomized and stratified clinical trial. They will be randomized to either continue with its usual high activity antiretroviral therapy (HAART) treatment or to receive 300 mg of Maraviroc every 12 hours plus its usual treatment. After 24 weeks, lymphocyte counts will be assessed, as well as safety, clinical progression, immunological profile of the patients and the potential benefit of Maraviroc for HIV+ cirrhotic patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* HIV infection
* Patients receiving HAART treatment for at least one year with a sustained viral load equal or below 200 copies/ml
* Viral load equal or below 200 copies/ml at the screening visit
* Discordant patients: patients without an increment over 50 copies /ml of CD4 lymphocytes during the last year
* Patients with an expected adherence to HIV treatment over 90% according to their physician.
* Signed informed consent form

Exclusion Criteria:

* Pregnancy or breast feeding or women planning pregnancy during the study duration
* Any contraindication to treatment with Maraviroc
* X4 tropism at inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)

PRIMARY OUTCOMES:
Median of CD4 counts change after 24 weeks | 24 weeks

SECONDARY OUTCOMES:
Immunological profile | 24 weeks
  Immunohistochemistry and flow cytometry techniques will be performed on peripheral blood to study immunological response to Maraviroc treatment
CD4 counts | 24 weeks
  Number of pacients with CD4 counts over 200 cells/mm3
Clinical progression | 24 weeks
  Progression to diseases classified as category C in CDC HIV guidelines; to other diseases or patient death

CONTACTS AND LOCATIONS:
Overall Officials: José Luis Blanco, MD, Principal Investigator — Hospital Clínic i Provincial
Locations (1):
- Hospital Clínic i Provincial, Barcelona, Barcelona, Spain